CLINICAL TRIAL: NCT05527210
Title: Prebiotic Treatment in People With Schizophrenia
Acronym: FOCIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Robert Buchanan, Chief, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HP-00102648; R61AT009990 (NIH)
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Prebiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Study Med (Active Comparator): Participants randomized to active study medication will mix 4g of powder prebiotic with water, 3 times a day for 12 weeks.
  Interventions: Dietary Supplement: Prebiotic
- Placebo (Placebo Comparator): Participants randomized to active study medication will mix 4g of powder placebo with water, 3 times a day for 12 weeks.
  Interventions: Dietary Supplement: Placebo Prebiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — Prebiotin® is a fine, white to slightly yellow powder, which is mixed into water and has a slightly sweet taste.
  Other Names: Prebiotin®
  Arms: Active Study Med
Dietary Supplement: Placebo Prebiotic — Placebo prebiotic mixed into water
  Other Names: maltodextrin
  Arms: Placebo

SUMMARY:
The proposed project is based on the observation that schizophrenia is characterized by a chronic pro-inflammatory state, which contributes to the severity of a number of the clinical manifestations of the illness, including cognitive impairments, the treatment of which represents a critically important unmet therapeutic need.

DETAILED DESCRIPTION:
The investigators hypothesize that the level of inflammation in people with schizophrenia can be reduced through the use of the prebiotic: Prebiotin®, an oligofructose-enriched inulin (OEI), to stimulate the activity of butyrate-producing bacteria and increase the production of butyrate, which has multiple anti-inflammatory properties. The investigators will confirm the effect of prebiotic administration on the biological signature and examine whether increased serum butyrate levels are associated with changes in cognitive performance (primary specific aim), symptoms, and metabolic measures; and the extent to which these associations are mediated by the anti-inflammatory properties of butyrate, including the ability of butyrate to decrease gut permeability and inhibit the production of pro-inflammatory cytokines, and/or changes in gut microbiota composition.

In a sample of participants with a DSM-5 diagnosis of schizophrenia or schizoaffective disorder, the investigators will conduct a 12-week, double-blind, placebo-controlled, randomized clinical trial to confirm the effect of prebiotic administration on the biological signature and examine whether increased serum butyrate levels are associated with changes in cognitive performance, symptoms, and metabolic measures; and the extent to which these associations are mediated by the anti-inflammatory properties of butyrate, including the ability of butyrate to decrease gut permeability and inhibit the production of pro-inflammatory cytokines, and/or changes in gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of schizophrenia or schizoaffective disorder;
2. Age 18-60 years;
3. Considered clinically stable by the treating psychiatrist;
4. Currently treated with an antipsychotic, with no dose changes in last 14 days;
5. Ability to participate in the informed consent process, as determined by a score of 10 or greater on the Evaluation to Sign Consent;
6. BMI ≤ 40

Exclusion Criteria:

1. Gastrointestinal disorders, including, but not limited to Crohn's Disease, Irritable Bowel Syndrome, Celiac Disease, whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol
2. Organic brain disorder, including cerebrovascular accident; epilepsy; traumatic brain injury, Loss of consciousness (LOC) for more than 30 minutes
3. Intellectual disability
4. Acute antibiotic use
5. Immune therapy within the last three months
6. Prebiotic or probiotic treatment within the last three months
7. Inability to understand English
8. Inability to cooperate with study procedures
9. Pregnant or lactation secondary to pregnancy
10. Participants who meet DSM 5 criteria for alcohol or substance misuse (except caffeine and nicotine) within the last 3 months will be excluded. Participants who meet DSM 5 criteria for marijuana misuse - mild will be included in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum butyrate levels | 12 weeks
  Number of participants with an increase in serum butyrate levels at 12 weeks.
Cognition | 12 weeks
  Number of participants with an increase in MCCB composite score at 12 weeks.
Incidence of Side Effects | 12 weeks
  Number of participants with an increased incidence of side effects at 12 weeks.

SECONDARY OUTCOMES:
Change in Affective Symptoms | 12 weeks
  Number of participants with an increase in affective symptoms at 12 weeks, measured by the Calgary Depression Scale (CDS).
Change in Positive Symptoms | 12 weeks
  Number of participants with an increase in positive symptoms at 12 weeks, measured by the Brief Psychiatric Rating Scale (BPRS).
Change in Negative Symptoms | 12 weeks
  Number of participants with an increase in negative symptoms at 12 weeks, measured by the • Scale for the Assessment of Negative Symptoms (SANS).
Changes in Serum Measurements | 12 weeks
  Number of participants with an increase in fasting levels of serum glucose, triglycerides, and/or cholesterol at 12 weeks.
Effects of Gut Composition | 12 weeks
  Number of participants with an increase in cytokine, gut permeability, or gut microbiota composition levels at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Buchanan, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Maryland Psyciatric Research Center, Catonsville, Maryland, United States